CLINICAL TRIAL: NCT01397370
Title: Double Blind, Placebo Controlled Dose Ranging Study for the Assessment of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Oral Doses of GLPG0492 in Healthy Subjects
Brief Title: Multiple Ascending Dose Study of GLPG0492 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: GLPG0492-CL-102; 2010-024039-18 (EudraCT Number)
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — 4-(4-(hydroxymethyl)-3-methyl-2,5-dioxo-4-phenylimidazolidin-1-yl)-2-(trifluoromethyl)benzonitrile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLPG0492 oral solution (Experimental): Multiple ascending doses once daily for 14 days, starting from 5 mg/day
  Interventions: Drug: GLPG0492
- Placebo oral solution (Placebo Comparator): Once daily dosing for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG0492 — Oral solution
  Arms: GLPG0492 oral solution
Drug: Placebo — Oral solution
  Arms: Placebo oral solution

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of multiple ascending oral doses (MAD) of GLPG0492 given to healthy subjects for 14 days compared to placebo, and to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of GLPG0492 after multiple oral administrations.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years
* body mass index (BMI) between 18-29.9 kg/m², inclusive.
* normal values of testosterone (2.49-8.36 ng/mL) and LH (1.7-8.6 U/L)

Exclusion Criteria:

* smoking
* drug or alcohol abuse
* hypersensitivity to any of the ingredients of the study drug

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of GLPG0492 in terms of adverse events, vital signs, ECG and abnormal lab tests in comparison with placebo | Up to 2 weeks after last treatment
  Occurrence of adverse events, vital signs, ECG and abnormal lab tests as a measure of safety and tolerability

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile and metabolism after single and multiple doses of GLPG0492 | Up to 2h hours after last treatment
  The plasma levels of GLPG0492 will be determined as a measure of pharmacokinetics, and the plasma and urine levels of GLPG0492 will be used for metabolism investigation
To assess whether GLPG0492 induces CYP450, a pharmacodynamic marker by measuring the ratio of β-OH-cortisol /cortisol in urine | Up to 24 hours after last treatment
  To assess the potential of daily doses of GLPG0492 to induce cytochrome P450(CYP3A4), a pharmacodynamic marker, by measurement of the ratio of β-OH-cortisol /cortisol in urine

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- Parexel Early Phase Clinical Unit, Berlin, Germany